CLINICAL TRIAL: NCT01359371
Title: Evaluation of Peer Telephone Cessation Counseling for Smokers
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: RRP 11-020
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Smoking
Keywords: Smoking Cessation; Telephone; Hospital Volunteers
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Peer telephone cessation counseling: The cohort is 131 veteran smokers who received the standard-of-care Tobacco Tactics intervention while in the hospital follow up volunteer peer telephone cessation counseling
  Interventions: Behavioral: Peer telephone cessation counseling

INTERVENTIONS:
Behavioral: Peer telephone cessation counseling — For Veterans who received the inpatient Tobacco Tactics intervention, trained volunteers initiated follow-up telephone cessation counseling at 2, 14, 21 and 60 days after in-patient discharge; three attempts were made per time point.
  Other Names: Tobacco Tactics

SUMMARY:
The purpose of this study is to evaluate the peer telephone cessation counseling that has been and continues to be implemented at the Ann Arbor VA as part of the Tobacco Tactics intervention.

DETAILED DESCRIPTION:
Background: As part of the nurse-administered Tobacco Tactics intervention, we developed a novel program to train veterans from Voluntary Services to provide peer telephone cessation counseling calls.

Objectives: The objective of this study is to conduct an in-depth evaluation of the volunteer peer telephone cessation counseling that has been implemented and continues to be implemented at the Ann Arbor Veterans Affairs (VA) hospital as part of the inpatient Tobacco Tactics intervention.

Methods: Using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework, this quasi-experimental study will collect both quantitative and qualitative data to evaluate the peer telephone cessation counseling component of the Tobacco Tactics intervention. The Reach of the program will be evaluated by determining differences in the demographics, health characteristics, and smoking characteristics of those who do and do not participate in the peer telephone cessation counseling. The Effectiveness of the program will be evaluated by determining if there were differences in quit rates between those that do and do not participate in the peer telephone cessation counseling. The Adoption and Implementation of the program will be evaluated by determining the satisfaction with the counseling, reasons for nonparticipation, the type and quality of counseling actually provided, and barriers and facilitators to implementing the counseling as perceived by staff. The Maintenance of the program will be evaluated by determining the estimated costs of implementing the peer telephone cessation counseling.

Impact: The Tobacco Use/Smoking Cessation goal of the VA Substance Use Disorders (SUD) Quality Enhancement Research Initiative (QUERI) is to develop, implement and evaluate cost-effective interventions for increasing access to and use of evidence-based smoking cessation treatment. Telephone counseling has been shown to be efficacious and teaching volunteer veterans to provide this service is an option that is likely to be cost effective. Hence, evaluating the peer cessation telephone counseling program at the Ann Arbor VA will provide valuable information as to whether or not the program is a viable option for wider scale dissemination.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria: veterans who received the Tobacco Tactics intervention as an inpatient in the hospital.

Exclusion Criteria:

* The exclusion criteria: veterans who are too ill or impaired to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatient veterans at the Ann Arbor VA
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia A. Duffy, PhD MS RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Duffy SA, Ewing LA, Louzon SA, Ronis DL, Jordan N, Harrod M. Evaluation and costs of volunteer telephone cessation follow-up counseling for Veteran smokers discharged from inpatient units: a quasi-experimental, mixed methods study. Tob Induc Dis. 2015 Feb 5;13(1):4. doi: 10.1186/s12971-015-0028-9. eCollection 2015. PMID 25674045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were provided with the Tobacco Tactics manual as part of their inpatient hospitalization were automatically referred to the volunteer telephone cessation counseling program.
Groups:
- Volunteer Telephone Cessation Counseling: The cohort is discharged veteran smokers who received the standard-of-care Tobacco Tactics intervention while in the hospital.
Period: Overall Study
Arm/Group | Volunteer Telephone Cessation Counseling
Started | 131
Completed | 131
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Volunteer Telephone Cessation Counseling: The cohort is discharged veteran smokers who received the standard-of-care Tobacco Tactics intervention while in the hospital an follow-up volunteer peer telephone counseling
Arm/Group | Volunteer Telephone Cessation Counseling
Number analyzed (Participants) | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 115
  More than one race | 0
  Unknown or Not Reported | 10

OUTCOME MEASURES:

1. Primary Outcome: Smoking Quit Rate by Number of Calls Received
Description: Smoking status around 60-days post-discharge (range 1 month to 5 months) was collected from electronic medical record text fields (smoked in the past 7 days-yes/no) or 60-day volunteer documentation (smoked in the last 24 hours-yes/no). When smoking status data was missing, participants were considered to be a smoker.
Time Frame: 7-day point prevalence self-reported smoking quit rate 60 days after discharge
Measure: Count of Participants; unit: Participants
Groups:
- Quit Rate With Low Participation in Counseling: Quit rate of those reached 0-1 times for peer telephone counseling.
- Quit Rate High Participation in Counseling: Quit rate of those reached 2-4 times for peer telephone cessation counseling.
Arm/Group | Quit Rate With Low Participation in Counseling | Quit Rate High Participation in Counseling
Number analyzed (Participants) | 25 | 106
Participants | 1 | 35
Statistical Analysis 1: Comparison: Quit Rate With Low Participation in Counseling vs Quit Rate High Participation in Counseling; Bivariate relationships between a patient's participation in the program and smoking status were calculated; Test type: Superiority; p < .01, Fisher Exact

2. Secondary Outcome: Characteristics of Participants Stratified by High vs. Low Participation 60 Days Post Discharge
Description: Demographics and health characteristics of those who had high participation (2-4 contacts) versus low (0 to 1 contacts) in the telephone counseling program (Reach) Row totals may vary due to missing data.
Time Frame: 60 days after discharge
Population: Row totals may vary due to missing data.
Measure: Number; unit: participants
Groups:
- High Participation: Reached 2-4 times for telephone counseling
- Low Participation: Reached 0-1 times for telephone counseling
Arm/Group | High Participation | Low Participation
Number analyzed (Participants) | 106 | 25
participants
  Male | 101 | 24
  Female | 5 | 1
  Non-Hispanic White | 94 | 21
  Other race/ethnicity | 11 | 4
  Married | 36 | 8
  Not Married | 69 | 17
  High School/GED or less | 59 | 13
  Some college or more | 45 | 11
  Employed | 18 | 7
  Unemployed | 87 | 18
  Comorbid lung disease yes | 39 | 2
  No comorbid lung disease | 67 | 23
  0-2 Comorbidities | 22 | 7
  3 or more comorbidities | 84 | 18
  Used tobacco past 7 days | 78 | 23
  No tobacco use past 7 days | 28 | 2
  Used tobacco last 24 hours | 71 | 24
  No tobacco use past 24 hours | 35 | 1
Statistical Analysis 1: Comparison: High Participation vs Low Participation; Test type: Other — T-tests, chi squares and Fishers exact tests were used to compare groups; p < .05, Chi-squared — This was just a sample description, so there was not adjustment for multiple comparisons; T-tests, chi squares and Fishers exact tests were used to compare groups
Statistical Analysis 2: Comparison: High Participation vs Low Participation; T-tests, chi squares and Fishers exact tests were used to compare groups; Test type: Other; p < .05, Chi-squared

3. Secondary Outcome: Participants' Attitudes About the Implementation of the Telephone Counseling
Description: Thirty-minute qualitative telephone interviews were conducted with Veteran smokers that participated in the volunteer peer telephone cessation counseling.
Time Frame: 60 days after discharge
Population: Of those surveyed, 25 agreed to qualitative phone interviews.
Measure: Count of Participants; unit: Participants
Groups:
- Interviews With Veterans About Satisfaction: 25 of the 131 Veteran smoker participants who received the standard-of-care Tobacco Tactics intervention while in the hospital and were interviewed about their satisfaction with the volunteer peer telephone cessation counseling.
Arm/Group | Interviews With Veterans About Satisfaction
Number analyzed (Participants) | 25
Participants
  Wanted to quit smoking | 19
  Liked the program in hospital | 9
  Calls were helpful/good/great | 23
  Liked that someone cared | 16
  Liked the number of calls | 14
  Would have liked more calls | 12
  Can't remember content of calls | 3
  Calls put quitting back in head | 3
  No difference in smoking after calls | 11
  Increased smoking after calls | 6
  Decreased smoking after calls | 4
  No suggestions for changes in calls | 18
  Increase number of calls | 6
  Make smoking medications more accessible | 5
  Provide more information on calls | 1

4. Secondary Outcome: Cost Per Quit of Volunteer Peer Telephone Counseling
Description: The primary cost component of the intervention is the cost of labor by providers to train the volunteers and enter volunteer documentation into the electronic medical record. These costs were estimated using VA salary and fringe benefit information obtained from the Financial Management System (FMS). Number of hours spent by the volunteers providing telephone counseling was also tracked. Other intervention costs included nominal supplies associated with training and the intervention. Because the volunteers made their telephone calls in an unused office, the cost of space was not included. Recruitment and other research-related costs were excluded. The average cost per quit is a mean, but is reported here as a number, as no measures of dispersion were available.
Time Frame: 60 days after discharge
Measure: Number; unit: dollars
Groups:
- Costs Per Quit of Peer Cessation Telephone Counseling: The cohort is 131 Veteran smokers who received the standard-of-care Tobacco Tactics intervention while in the hospital and were interviewed about their satisfaction with peer cessation telephone counseling and 4 peer telephone counselors.
Arm/Group | Costs Per Quit of Peer Cessation Telephone Counseling
Number analyzed (Participants) | 131
dollars | 92

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Volunteer Telephone Cessation Counseling
Serious Adverse Events (participants affected / at risk) | 0/131
Other Adverse Events (participants affected / at risk) | 0/131

LIMITATIONS AND CAVEATS:
Quasiexperimental study with no control group. Potential selection bias. Quit rates were not cotinine-verified. Small sample size. One site4 study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes